CLINICAL TRIAL: NCT06052943
Title: Family-Inclusive Lifestyle Intervention for Teenagers in Rural Colorado
Brief Title: Health Without Barriers/Salud Sin Barreras
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: Colorado State University Extension-La Plata County (Unknown); United States Department of Agriculture (USDA) (U.S. Federal Agency); University of Colorado, Denver (Other); Colorado Health Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1883
Record Dates: First submitted 2023-08-25; First posted 2023-09-25 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Mental Health Wellness; Family Research; Lifestyle Risk Reduction
MeSH Terms: conditions — Risk Reduction Behavior | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health without Barriers/ Salud Sin Barreras (Experimental): Health Without Barriers/Salud Sin Barreras is 12-session community-delivered, family-based lifestyle intervention to reduction the risk of for chronic diseases (i.e., T2D) in adolescence and to improve whole family health and wellness. The program is based upon a lifestyle intervention called the Healthy Living Program (HeLP), which includes 6 weekly 2 hour nutrition/cooking sessions through Cooking Matters and 6 weekly 2 hour Multidisciplinary Sessions that include parent education, a teen and sibling (ages 6-10 years) group physical fitness class, preschool curriculum for children 2-5 years of age, and a teen mindfulness curriculum called Learning 2 BREATHE. Health Without Barriers/Salud Sin Barreras has been tailored for adolescents at risk for depression and chronic diseases (i.e., T2D) in Southwest Colorado based on community input.
  Interventions: Behavioral: Mindfulness-Based Intervention; Behavioral: Parent Education; Behavioral: Physical Activity; Behavioral: Brief Mindfulness Intervention for Parents; Behavioral: Preschool Curriculum; Behavioral: Cooking Matters

INTERVENTIONS:
Behavioral: Mindfulness-Based Intervention — Learning 2 BREATHE (L2B) is an evidence based curriculum for adolescents. L2B in this program consists of 6 sessions of approximately 1 hour per session. In between sessions, participants are asked to practice brief mindfulness skills individually.
  Other Names: Learning 2 BREATHE
Behavioral: Parent Education — The parent education curriculum includes 3 modules: 1) family support/parenting, 2) nutrition and 3) physical activity. The parents set weekly goals to implement the parent education lessons into everyday living.
Behavioral: Physical Activity — Combines aerobic and resistance training though game play.
Behavioral: Brief Mindfulness Intervention for Parents — Parent-based mindfulness education based on the Learning to BREATHE curriculum.
Behavioral: Preschool Curriculum — Preschool age children learn about and try new foods.
Behavioral: Cooking Matters — Nutrition education and hands-on cooking lessons for the whole family

SUMMARY:
The goal of this study is to address a key health inequity - lack of community access to evidence-based programs to prevent chronic health conditions (e.g., Type 2 Diabetes) - by tailoring and delivering a family-based lifestyle and stress management intervention, Health Without Barriers/Salud Sin Barreras, for adolescents and their families living in rural Southwest Colorado. The intervention is a lifestyle program that addresses healthy lifestyle habits within the family context to support adolescent mental health (mindfulness intervention) and healthy weight (physical activity, nutrition, and parent education).

DETAILED DESCRIPTION:
Health Without Barriers/Salud Sin Barreras is a 12-session community-delivered, family-based lifestyle intervention for health promotion and reduction of risk for chronic diseases like T2D. The program is delivered over 6 weeks and includes family education/parent training, adolescent physical activity, mindfulness-based stress reduction training for adolescents, family meals, and family cooking/meal preparation. The goal is to deliver the program to up to 175 participants and their families over the course of 5 years (2022-2027). The program content and delivery/implementation processes already have been adapted based on information obtained through adolescent and parent interviews and community member voices though a 9-month community research collaboration. The investigators will gather new, additional information from program participants and stakeholders to continue to tailor the curriculum content and program processes. The investigators will do this iteratively using feedback collected during and in the wake of each cohort until thematic saturation is achieved (anticipated to be ~3 cohorts) and until the community-research partnership group has obtained program optimization for families in Southwest Colorado. Further, the investigators will conduct program evaluations of the adapted Health Without Barriers/Salud Sin Barreras program on changes in a range of indicators of mental/physical health and health behaviors in adolescents.

ELIGIBILITY:
Inclusion Criteria:

Families must have at least 1 teen that is between the ages of 11-19 years old and reside in La Plata, Montezuma, or Archuleta Counties.

Exclusion Criteria:

* Participants will not take part in the program and/or research activities if they have a medical and/or psychological/behavioral condition that, in the opinion of the Colorado State University/Extension program team, could interfere with safety for themselves or others or interfere with the capability of the participant or other participants to potentially benefit from the program (e.g., severe emotional-behavioral disturbance, inability to follow facilitator directions) .
* Parents/guardians will not take part in the program and/or research activities if they have a medical and/or psychological/behavioral condition that, in the opinion of the Colorado State University/Extension program team, could interfere with safety for themselves or others or interfere with the capability of their family or other participating families to potentially benefit from the program (e.g., using drugs or alcohol or under the use of drugs/alcohol during program sessions, aggressive or inappropriate behavior toward other participants).

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 175 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Treatment Acceptability: Questionnaire | 6 weeks
  Participants rate and comment on each component of the program (i.e. Cooking Matters, parent sessions, physical fitness sessions, Learning 2 BREATHE, dinners) separately. Questions include topics about how supported individuals felt during the program, the helpfulness of the facilitators, the perceived benefits of program participation, and their overall experience participating in the program. This questionnaire will only be completed one time at the post-program follow-up.
Intervention Acceptability: Qualitative Themes | 6 weeks
  Themes indicative of acceptability of intervention obtained from qualitative analysis of participant and parent focus-groups at post-intervention.

SECONDARY OUTCOMES:
Emotion regulation | 1 year
  Difficulties in Emotion Regulation Scale-Short Form (18 items), measures non-acceptance of emotional responses, difficulty engaging in goal-directed behavior, impulse control difficulties, lack of emotional awareness, limited access to emotion regulation strategies, and lack of emotional clarity.
Eating behavior | 1 year
  Reward-Based Eating Drive Scale (REDS), a reliable/valid survey instrument of hedonic eating
24-hour dietary intake | 1 year
  NIH Automated Self-Administered 24-Hour (ASA24) Dietary Assessment Tool in order to assess dietary intake, including total energy intake, macronutrients, fruits/vegetable consumption, and overall quality of diet.
Physical activity- engagement | 1 year
  NIH Patient-Reported Outcomes Measurement Information System (PROMIS): Pediatric Physical Activity - Short Form, measures the number of times an individual engaged in different types of physical activity in the past 7 days.
Physical activity- self-confidence | 1 year
  Exercise Self-Efficacy Scale, measures an individual's beliefs in their ability to continue exercising on a three time per week basis at moderate intensities for 40 or more minutes per session in the future.
Sleep disturbance | 1 year
  4-item PROMIS Pediatric Sleep Disturbance Short Form, measures the frequency an individual experienced disturbed sleep in the past 7 days.
Cardiometabolic health | 1 year
  Finger prick by lancet is used to analyze HbA1c, HDL/LDL cholesterol, and triglycerides.
Daily glucose patterns | 1 year
  Continuous glucose monitoring is used to describe average daily glucose, peak glucose, SD, and mean amplitude of glycemic excursions.
Blood Pressure | 1 year
  Blood pressure assessed via digital blood pressure monitor.
Height and Weight | 1 year
  Weight will be measured via scale and height via stadiometer. These measures are used to calculate BMI percentile. Fasted weight measurement is taken via scale and is optional for participants.
Body Composition Measurement | 1 year
  Body composition is measured using bioelectrical impedance analysis (BIA). BIA is performed using a validated bioelectrical impedance scale.
Activity Monitoring | 1 year
  Participants will be fitted with a ActiGraph GT9X Link and asked to wear the device for 7 days.
Sleep Monitoring | 1 year
  Participants will be fitted with a ActiGraph GT9X Link and asked to wear the device for 7 days.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Colorado State University Extension, Durango, Colorado
  - Colorado State University, Fort Collins, Colorado

IPD SHARING:
Plan to Share IPD: No